CLINICAL TRIAL: NCT05751772
Title: Disease and Medication Knowledge Improvement: A Swiss Single-center Randomized Controlled Trial With Heart Failure Inpatients
Brief Title: Improving Knowledge in Heart Failure Inpatient With Therapeutic Education
Acronym: EDUC-IC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting and lack of resources
Sponsor: University Hospital, Geneva (Other)
Collaborators: Vifor Pharma (Industry); Labatec Pharma SA (Industry); Bayer (Industry); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Mégane Jermini, Hospital and Clinical Pharmacist, pharmD, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-00731
Record Dates: First submitted 2022-11-04; First posted 2023-03-02 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Heart Failure; With Decompensation; Pharmacist-Patient Relations; Medication Adherence; Knowledge, Attitudes, Practice
Keywords: patient therapeutic education; clinical pharmacy; pharmaceutical care
MeSH Terms: conditions — Heart Failure; Medication Adherence; Behavior

STUDY DESIGN:
Intervention Model Description: Single-center randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Patient therapeutic education" group (Experimental): The intervention group will benefit from a pharmacist-led therapeutic education intervention on the knowledge of hospitalized heart failure patients and usual hospital care (medical and nursing care)
  Interventions: Other: Patient therapeutic education
- "Usual hospital care" group (No Intervention): The control group do only benefit from the usual hospital care (any medical and nursing care giving to an acute heart failure inpatient) and won't benefit from the pharmacist's educational intervention.

INTERVENTIONS:
Other: Patient therapeutic education — The pharmacist-led therapeutic education intervention on the knowledge of hospitalized heart failure patients is made by a clinical pharmacist and includes:
  1. Targeted education on patient needs related to heart failure, heart failure medications and self-care;
  2. a pre-discharge interview to consolidate key teaching messages and prepare the patient for their discharge treatment plan;
  3. a telephone call the week of discharge to ensure pharmaceutical follow-up between hospital care and return home (continuity of care, transition of care).
  Other Names: inpatient therapeutic education interview and outpatient pharmaceutical follow-up
  Arms: "Patient therapeutic education" group

SUMMARY:
The objective is to evaluate the impact of a pharmacist-led therapeutic education intervention on the knowledge of hospitalized heart failure patients. The knowledge score on heart failure disease and medications will be compared between two groups one month after hospitalization. The intervention group will receive a therapeutic education intervention and usual hospital care and the control group will receive only usual hospital care.

DETAILED DESCRIPTION:
Heart failure patients are at risk of decompensation of their disease and frequent hospitalizations. Poor adherence to their treatment may be the cause. By improving the knowledge of hospitalized heart failure patients about their disease and their medications, it is expected that these patients will adhere better to their heart failure drug therapy and benefit from a better effectiveness of their treatment. This could promote an improvement in their quality of life, a decrease in their risk of disease complications and even an increase in their life expectancy.

The objective of this research project is to deploy a therapeutic teaching intervention at the bedside of decompensated and hospitalized heart failure patients, associated with follow-up by the pharmacist at discharge from the hospital, and to measure its impact on knowledge change (primary endpoint), on their beliefs about medications, on their therapeutic adherence, and on the consumption of unplanned care such as rehospitalizations and emergency room visits (secondary endpoints).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in the Department of General Internal Medicine or Cardiology for decompensated heart failure with lowered left ventricular ejection fraction (LVEF) (≤40%) from any cause or mildly lowered LVEF (41-49%) with the presence of heart failure-specific drug therapy
* Stability of the patient's clinical condition
* ≥ 2 heart failure medications
* ≥18 years
* Full capacity of discernment
* Absence of cognitive impairment
* Ability to speak, understand and read in French
* Get a personal telephone
* Consent form signed by the participant

Exclusion Criteria:

* Inability to follow study procedures
* Institutionalized persons
* Asylum seekers, homeless people, prisoners
* Incapacity of judgment and discernment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Change in knowledge score | at the baseline time (zero time), immediately after therapeutic education intervention and 30 days after hospital discharge
  Patients' level of knowledge about their disease and heart failure medications before the educational pharmaceutical intervention (pre-test) and immediately after the intervention (post-test n° 1) for the intervention group , as well as at 1 month after hospital discharge (post-test n°2) for the intervention and control group. It will be measured by means of a 17-question questionnaire specifically developed for this project. This level is valued by a minimum score of 0 points and a maximum of 17 points. Higher score means a better level of knowledge. The positive difference between pre-test and post-tes means an increase in knowledge and a negative difference means a decrease in knowledge.

SECONDARY OUTCOMES:
Change in Beliefs about medicines Score | at the baseline time (zero time),30 days after hospital discharge
  Beliefs about medicines will be measured via the specific Beliefs about Medicines Questionnaire (BMQs) score at baseline time (at the inclusion time)(pretest) and at 1 month after hospital discharge (post-test) in both groups.
  Scores range from 5 to 25 points for both subscales. The higher the score for the specific need, the more it means that the patient has a strong perception that he needs the drugs to be healthy and live. For specific concerns, the higher the score, the more the patient is concerned about a potential negative effect of taking the medication. A third score can be calculated by subtracting specific concerns from specific needs. This gives a score of -20 to +20. A positive value means that the need for the treatment exceeds the concerns of taking it.
Change in Medication Adherence Score | at the baseline time (zero time),30 days after hospital discharge
  Adherence will be assessed with the Three Item Self Report Scale at baseline time (at the inclusion time) (pre-test) and at 1 month after hospital discharge (post-test) in both groups.
  This questionnaire consists of 3 questions; one which evaluates the number of days of forgetting to take medication over the last month, one which evaluates the frequency of taking medication according to medical prescription and the third which makes it possible to measure the level of competence in the correct taking of medication that takes ownership of the patient. Responses are converted on a scale of 0 to 100 (0 is the lowest adherence and 100 the highest). An average of the three answers is used to assign the adhesion score. Higher the score is, better the adherence is.
Level of satisfaction on therapeutic education | immediately after therapeutic education intervention
  Patient satisfaction will be assessed using a 13-questions questionnaire specifically developed for this project, after the education interview to assess the usefulness and quality of the teaching intervention. There is no score related to the questionnaire.
  This qualitative assessment will allow us to determine whether this new intervention should be continued and to identify its strengths and weaknesses.
Rehospitalization or emergency room visits | 30 days after hospital discharge
  The rate of rehospitalization or emergency room visits will be evaluated during the telephone call made by a research assistant at D30 post hospital discharge. The cause of hospitalization will be determined by means of the computerized hospital patient file if he is rehospitalized at the university hospital of Geneva (HUG) or directly to the patient (or his attending physician depending) if he is hospitalized in another hospital. It is interesting to assess whether the patient consumed unplanned care and whether it was related to instability of his heart failure.
Death at 1 month after discharge | 30 days after hospital discharge
  The mortality rate will be assessed in both groups. This information can be collected from the participants' computerized patient records if mentioned or from the participants' relatives or attending physician.
Patient experiment and feeling after discharge | 7 days after hospital discharge
  The patient's experience and feelings upon returning home will be assessed during a telephone call between D3 and D7 after the patient's discharge from the hospital with open questions (no validated questionnaire is used). The objective will be to identify the patient's needs, their feelings about going home, what they liked, what they missed to readjust the counseling to the patient.
CardioMeds app usability | 30 days after hospital discharge
  Use and usability of the mobile smartphone application (CardioMeds® ) will be explored by the research assistant during the telephone call at D30 post hospital discharge using a validated standardized questionnaire (System Usability Scale = SUS).
  SUS gives a single score representing a measure composite of the general user-friendliness of the studied service.
  The score ranges from 0 to 100.It is generally considered that a score is "good" from 75, fair or fair between 50 and 75. A score below 50 reveals major problems in terms of customer satisfaction.
Self-Care of Heart Failure Index | 30 days after hospital discharge
  Self-care skills of patients using CardioMeds® will be explored using a validated score, the Self-Care of Heart Failure Index composed of 22 questions to measure the effect of this application on patients' level of empowerment in their care. The scale is subdivided in three measurement : maintenance score, management score and self-care confidence score. Each scale score is standardized to a 0 to 100 range. A score of ≥70 can be used as the cut-point to judge self-care adequacy,
Level of satisfaction on global pharmaceutical care | 30 days after hospital discharge
  This second satisfaction questionnaire consisting of 8 questions specifically developed for this project, will be sent at 1 month after hospital discharge to assess the patient's overall satisfaction with the pharmaceutical care follow-up provided. There is no score related to the questionnaire.
  This qualitative assessment will allow us to determine whether the hospital pharmaceutical care

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Bonnabry, Professor, Study Director — University of Geneva
Locations (1):
- University Hospital of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (original data sets) that underlie the results reported in published articles, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Start immediately following publication. No end date.
Access Criteria: With whom? Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  For what type of analysis? For individual participant data meta-analysis.
  How to access to available data? Proposals should be directed to megane.jermini@hcuge.ch or megane.jermini@gmail.com. To gain access, data requestors will need to sign a data access agreement. Data are available in University of Geneva's data warehouse (Yareta data depository) but without investigator support other than deposited metadata.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT05751772/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT05751772/ICF_001.pdf